CLINICAL TRIAL: NCT00056667
Title: Relaxation Response, Somatic Style and Rheumatoid Arthritis
Brief Title: Relaxation Response Training for the Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Arthur Joseph Barsky III,M.D., Vice Chair for Research, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AR047014 (NIH); R01AR047014 (NIH); NIAMS-088
Record Dates: First submitted 2003-03-20; First posted 2003-03-24 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Treatment; Pain; Relaxation Response; Cognitive Behavioral Therapy
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CBT plus relaxation response (Experimental): Participants will receive cognitive behavioral therapy plus relaxation response training
  Interventions: Behavioral: Relaxation response and cognitive behavioral therapy
- Relaxation Response (Active Comparator): Participants will receive relaxation response training
  Interventions: Behavioral: Relaxation response
- Education (Placebo Comparator): Participants will receive rheumatoid arthritis education
  Interventions: Other: RA education

INTERVENTIONS:
Behavioral: Relaxation response and cognitive behavioral therapy — The cognitive behavioral therapy program wwill incorporate relaxation training, a modified version of the RA treatment program developed by Bradley et al (1987) and shown to be effective. The cognitive behavioral techniques include problem solving, relabeling, enhanced awareness of pain behaviors, and attention refocusing. The RR component includes instruction in diaphragmatic breathing along with progressive skeletal muscle relaxation. The intervention will be modified from the original program in that neither biofeedback training nor participation of family members will be included. Consequently, the number of weekly group sessions will be reduced from 14 to 12. Homework will be given at the end of each session, to be completed and brought in for review to the next session.
  Other Names: RRCBT
  Arms: CBT plus relaxation response
Behavioral: Relaxation response — The relaxation response (RR) consists of a set of integrated physiological changes elicited when a participant engages in the repetitive mental action of focusing on a word, phrase, or image, while passively ignoring distracting thoughts. These changes include decreased oxygen consumption, heart rate, arterial blood pressure, respiratory rate, and arterial blood lactate, along with slight increases in skeletal muscle blood flow. The long-term physiologic changes of participants eliciting the relaxation response are consistent with reduced norepinephrine end organ responsivity. These latter changes provide a plausible psychophysiological mechanism for longer-term actions of the RR.
  Other Names: RR
  Arms: Relaxation Response
Other: RA education — RA education programs have been widely used to supplement routine medical care. They have been found to be of modest benefit, particularly in terms of knowledge about the condition and its treatment. The long-term effects on pain and level of function are less. When used as an attention control, such educational programs have been found to be as credible and as well attended as the active experimental treatment (Professor Francis Keefe, Personal Communication). In this study, patients randomized to the control condition will receive 8 weekly sessions of RA education, in groups of 6-10 patients each, using portions of the Arthritis Self-Management Program and incorporating printed and videotaped materials available from the Arthritis Foundation.
  Arms: Education

SUMMARY:
This study will evaluate the relative effectiveness of Relaxation Response (RR) training for the treatment of rheumatoid arthritis (RA). The study will compare RR training to RR training with cognitive behavioral therapy and to a standard RA education program.

DETAILED DESCRIPTION:
RR training is a part of most multi-component psychosocial therapies for RA. RR training may decrease perceived psychosocial stress and autonomic tone, which in turn diminishes pain and the anticipatory anxiety associated with pain. RR training involves learning relaxation techniques which include diaphragmatic breathing, progressive skeletal muscle relaxation, and the induction of a state of focused attention on a chosen word, phrase, or image.

In clinical practice, RR training is generally administered as one component of RA therapy. In this study, the effectiveness of RR training will be evaluated when RR training is administered alone and in combination with a cognitive behavioral therapy program. The cognitive behavior techniques include problem solving, relabeling, enhanced awareness of pain behaviors, and attention refocusing. The effectiveness of RR training will be evaluated in comparison to standard RA education that includes topics such as the nature of RA disease, medical therapies, physical activities, nutrition, and pain mechanisms.

After a baseline assessment of health beliefs, RA severity, social support, and psychological distress, patients will be randomized to one of three study arms. Patients in Arm A will complete six individualized weekly RR training sessions. Patients will receive a 20-minute audiotape to guide them through the exercise; they are asked to practice 5 to 7 times per week. Patients in Arm B will learn cognitive behavioral and RR techniques during eight weekly sessions. Patients in Arm C will receive standard RA education. After the initial training, all patients will be followed up with monthly telephone conversations for 4 months. Patients will have follow-up study visits at Months 6 and 12. Follow-up study visits include a medical interview, physical exam, and blood tests.

ELIGIBILITY:
Inclusion criteria

* RA as defined by the American College of Rheumatology
* English literacy and fluency

Exclusion criteria

* Major medical condition or illness which limits life expectancy or results in severe symptoms or functional disability (Duke Severity of Illness score > 0.85)
* Fibromyalgia
* Received or currently receiving psychosocial treatment for RA
* Unavailability for Month 12 follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2001-07; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Somatic symptoms as assessed by the Rheumatoid Arthritis Symptom Questionnaire | 12 months

SECONDARY OUTCOMES:
Role impairment and functional status as assessed with the Functional Status Questionnaire | 12 months
Medical care utilization as assessed with the hospital's automated encounter database | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Arthur J. Barsky, MD, Principal Investigator — Brigham & Women's Hospital, Boston, MA
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Barsky AJ, Ahern DK, Orav EJ, Nestoriuc Y, Liang MH, Berman IT, Kingsbury JR, Sy JT, Wilk KG. A randomized trial of three psychosocial treatments for the symptoms of rheumatoid arthritis. Semin Arthritis Rheum. 2010 Dec;40(3):222-32. doi: 10.1016/j.semarthrit.2010.04.001. PMID 20621334